CLINICAL TRIAL: NCT01103726
Title: Evaluation Of Regional Glucose Metabolism In Striatum As Measured By [18f]-Fluorodeoxyglucose Positron Emission Tomography Following Single Oral Dose Administration Of PF-02545920 In Healthy Subjects
Brief Title: Evaluation Of Striatal Glucose Metabolism With Positron Emission Tomography Following PF-02545920 In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: A8241013
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Healthy
Keywords: FDG-PET; regional cerebral glucose metabolism; striatum; PDE10 inhibitor
MeSH Terms: interventions — 2-((4-(1-methyl-4-pyridin-4-yl-1H-pyrazol-3-yl)phenoxy)methyl)quinoline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stage 1 (Experimental)
  Interventions: Drug: PF-02545920; Drug: placebo
- Stage 2 (Experimental)
  Interventions: Drug: PF-02545920; Drug: Placebo

INTERVENTIONS:
Drug: PF-02545920 — 1 and 5 mg tablets, 6 mg single dose
  Arms: Stage 1
Drug: placebo — matching placebo tablets, single dose
  Arms: Stage 1
Drug: PF-02545920 — 1 mg tablets, 3 mg single dose
  Arms: Stage 2
Drug: PF-02545920 — 5 mg tablets, 15 mg single dose
  Arms: Stage 2
Drug: Placebo — matching placebo tablets, single dose
  Arms: Stage 2

SUMMARY:
We hypothesize that PF-02545920 will increase glucose metabolism in a part of the brain called the striatum.

ELIGIBILITY:
Inclusion Criteria:

* Healthy right-handed male and female subjects between the ages of 18 and 55 years, inclusive
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs)
* An informed consent document signed and dated by the subject
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

* Women of reproductive potential
* History of agranulocytosis or movement disorder
* Positron Emission Tomography (PET) or Magnetic Resonance Imaging (MRI) contraindications

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2010-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Glucose metabolic rates in striatum using standard Region of Interest (ROI) analysis method. | Stage 1: Day 1, 8. Stage 2: Day 1, 8, 15.

SECONDARY OUTCOMES:
Whole brain glucose metabolic rate. | Stage 1: Day 1, 8. Stage 2: Day 1, 8, 15.
Relative glucose metabolic rate in striatum. | Stage 1: Day 1, 8. Stage 2: Day 1, 8, 15.
Glucose metabolic rate in striatal subregions: putamen and caudate nucleus. | Stage 1: Day 1, 8. Stage 2: Day 1, 8, 15.
Relative glucose metabolic rate in striatal subregions: putamen and caudate nucleus. | Stage 1: Day 1, 8. Stage 2: Day 1, 8, 15.
Glucose metabolic rate in striatum determined using data-driven ROI analysis method. | Stage 1: Day 1, 8. Stage 2: Day 1, 8, 15.
Relative glucose metabolic rate in striatum determined using data-driven ROI analysis method. | Stage 1: Day 1, 8. Stage 2: Day 1, 8, 15.
Effect size comparison between standard ROI and data-driven ROI analysis methods using both regional glucose metabolic rate and relative regional glucose metabolic rate. | Stage 1: Day 1, 8. Stage 2: Day 1, 8, 15.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8241013&StudyName=Evaluation%20Of%20Striatal%20Glucose%20Metabolism%20With%20Positron%20Emission%20Tomography%20Following%20PF-02545920%20In%20Healthy%20Subjects